CLINICAL TRIAL: NCT03839420
Title: Prospective Randomized Clinical Trial Comparing Early Rotation of Two Extended Depth of Focus Intraocular Lenses
Brief Title: To Compare Early Rotation of Two Extended Depth of Focus Intraocular Lenses
Acronym: VENUStoric
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carl Zeiss Meditec AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 929MP BER-401-18
Record Dates: First submitted 2019-02-01; First posted 2019-02-15 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Intervention Model Description: comparative randomized trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CZM IOL (Experimental)
  Interventions: Device: CZM IOL
- Competitor IOL (Active Comparator)
  Interventions: Device: Competitor IOL

INTERVENTIONS:
Device: CZM IOL — implantation of CZM IOL
  Arms: CZM IOL
Device: Competitor IOL — implantation of Competitor IOL
  Arms: Competitor IOL

SUMMARY:
To demonstrate that the Carl Zeiss Meditec (CZM) Extended depth of focus (EDOF) Intraocular lens (IOL) is superior to the competitor EDOF IOL with respect to Rotational Stability.

ELIGIBILITY:
Inclusion Criteria:

1. Patient informed of the consequences and constraints of the Clinical Investigational Plan and who has given his/her written informed consent
2. Patients of any gender, aged 18 or older
3. Assured follow-up examinations
4. Healthy eyes with clinically significant age related cataract requiring surgical treatment
5. Corrected distance visual acuity projected to be better than 0.2 logMAR after the cataract surgery, as determined by Investigator's medical judgment
6. Uni- and/or bilaterally regular corneal astigmatism ≥ 1.0 D and ≤ 3.0 D (confirmed by topography measurement)

8. Cataract density compatible with biometry measurement

Exclusion Criteria:

1. Patients unable to meet the limitations of the Clinical Investigational Plan or likely of non-cooperation during the trial
2. Patients whose freedom is impaired by administrative or legal order
3. Current participation in another drug or device investigation that affects patients vision
4. Ocular disorders, other than cataract, that could potentially cause future acuity loss
5. Have atonic pupil or physiologically small pupil (unable to dilate to at least 5 mm)
6. Any anterior segment pathology that could significantly affect outcomes (e.g. chronic or recurrent uveitis, iritis, aniridia, rubeosis iridis, etc.)
7. Abnormal corneal findings in either eye (e.g. keratoconus, pellucid marginal degeneration, or irregular astigmatism, clinically significant corneal membrane dystrophies)
8. Any condition in the study eye that could affect IOL stability (e.g. zonular dialysis, evident zonular weakness or dehiscence, Floppy iris syndrome etc.)
9. History of any clinically significant retinal pathology or ocular diagnosis (e.g. diabetic retinopathy, ischemic diseases, macular degeneration, retinal detachment, optic neuropathy optic nerve atrophy, amblyopia, strabismus, microphthalmus, epiretinal membrane, Choroidal hemorrhage etc.) in the study eyes that could alter or limit final postoperative visual prognosis
10. Pseudoexfoliation syndrome (according to investigator decision)
11. Pathologic miosis or Pharmacotherapy with miotic agent
12. Irregular astigmatism / Keratoconus
13. Uncontrolled glaucoma or IOP higher than 24mmHg under ocular hypertension treatment.
14. All kind of infections (acute ocular disease, external / internal infection, systemic infection)
15. Traumatic cataract
16. Monophthalmic patient
17. Patients, who are unable to fixate for a longer time, e.g. strabismus, nystagmus
18. Patient expected to require retinal laser treatment before the end of the last follow-up examination
19. Patient expected to require refractive laser treatment / refractive laser touch-up before the end of the last follow-up examination
20. Previous intraocular and corneal / refractive surgery
21. Current Systemic or ocular pharmacotherapy that effects patients vision (according to investigator decision)
22. Dementia
23. Previous use of cytotoxic drugs or total body irradiation within last 2 years
24. Any other pathology or condition presenting, according to the investigator opinion, a risk for the patient
25. Pregnancy and / or lactation period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2020-10-04 (Actual); Study Completion 2021-02-17 (Actual)

PRIMARY OUTCOMES:
IOL axis | Immediately after the surgery
  IOL axis will be analyzed based on images.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinikum Freiburg, Freiburg im Breisgau, Germany

IPD SHARING:
Plan to Share IPD: No